CLINICAL TRIAL: NCT02429882
Title: A Randomized, Double-blind, Placebo-controlled Study With an Open Label Extension to Evaluate the Safety and Efficacy of Brodalumab in Subjects With Axial Spondyloarthritis
Brief Title: Study of Efficacy and Safety of Brodalumab Compared With Placebo in Subjects With Axial Spondyloarthritis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Per Amgen's decision to discontinue co-development and co-commercialization of brodalumab, study is being cancelled/closed.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20101228; 2014-003701-15 (EudraCT Number)
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Axial Spondyloarthritis
Keywords: Ankylosing Spondyloarthritis; non-radiographic axial spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing; Non-Radiographic Axial Spondyloarthritis | interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brodalumab (Experimental)
  Interventions: Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Brodalumab 210 mg

INTERVENTIONS:
Drug: Brodalumab 210 mg — 210 mg brodalumab will be administered subcutaneously
  Arms: Placebo
Drug: Placebo — Placebo will be administered subcutaneously
  Arms: Brodalumab

SUMMARY:
The purpose of this study is to assess the safety and efficacy of brodalumab compared with placebo in participants with axial spondyloarthritis. Subjects will be randomized in a 1:1 ratio to brodalumab or placebo for the first part of the study. Subjects will then receive open label brodalumab for the remainder of the study. The entire study will be 312 weeks in duration for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Subject fulfills the ASAS classification criteria of axial spondyloarthritis (except Crohn's disease criterion) for > 3 months with age of onset < 45 years of age
* Subject has Bath Ankylosing Spondylitis DIsease Activity Index (BASDAI) score greater than or equal to 4 at screening and baseline
* Subject has spinal pain score (BASDAI question #2) greater than or equal to 4 at screening and baseline
* Subject has had adequate therapeutic trial (at least 4 weeks) of greater than or equal to 2 non-steroidal anti-inflammatory drgs (NSAIDs) at the maximum recommended dose unless contraindicated or subject is intolerant
* For subjects receiving non-biologic DMARDS subject has received treatment for greater than or equal to 3 months with a stable doe for greater than or equal to 4 weeks prior to initiation of IM
* For subjects receiving oral corticosteroids: the subject must be on a stable dose (not to exceed the equivalent of 10 mg of prednisone per day) for equal to or greater than 4 weeks prior to initiation of IMP

Exclusion Criteria:

* Complete ankylosis (fusion) of the spine; Subject has a positive test for tuberculosis
* Subject has a planned surgical intervention between baeline and week 16
* Subject has an active infection or history of infections as follows (any active infection for which systemic anti-infectives were used within 28 day prior to the first MP dose
* A serious infection, defined as requiring hospitalization or intravenous anti-infectives within 8 weeks prior to the first IMP dose
* Recurrent or chronic infections or other active infection that, in the opinion ofthe investigator might cause this study to be detrimental to the subject)
* Subject has active Crohn's disease or a history of Crohn's disease
* Subject has active ulcerative colitis requiring daily use of immunosuppressive therapy
* Subject has had active fibromyalgia within the past 12 months
* Subject has a prior history of greater than 1 anti-TNF therapy for ankylosing spondylitis
* Subject has used commercially available or investigational biologic therapies for ankylosing spondylitis as follows

  * Anti-tumor necrosis factor (TNF) therapy as follows: within 1 month prior to IMP initiation for etanercept and within 2 months prior to IMP initiation for other anti-TNF agents.
  * Other experimental or commercially available biologic therapies for ankylosing spondylitis within 3 months prior to IMP initiation
  * Anti-IL17 biologics (eg, brodalumab, secukinumab, ixekizumab) or anti-IL12/IL23 biologic therapy (eg, ustekinumab, briakinumab) at any time
  * Rituximab at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Assessment of SpondyloArthritis international Society (ASAS) | Week 16
  Achievement of Assessment of SpondyloArthritis international Society (ASAS) 20 response at week 16

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (3):
  - Research Site, Scottsdale, Arizona
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Duncansville, Pennsylvania
- Research Site, Winnipeg, Manitoba, Canada

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com